CLINICAL TRIAL: NCT01158755
Title: Comparison of Intensive Treatment Regimens and Standard Treatment Regimen for Tuberculous Meningitis: Pharmacokinetics, Pharmacodynamics and Tolerability Study
Brief Title: Intensified Treatment Regimens for TB Meningitis: PK, PD and Tolerability Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Ahmad Rizal Ganiem, MD, Universitas Padjadjaran
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: TB-201006.01
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Meningitis, Tuberculous; Pharmacokinetics; Pharmacodynamics; Tolerability
Keywords: Meningitis, tuberculous; Intensified Regimen; PK/PD and tolerability; Outcome
MeSH Terms: conditions — Tuberculosis, Meningeal | interventions — Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard dose rifampisin (Active Comparator): Subjects in this arm receive 450 mg rifampicin orally.
  In accordance with national TB treatment standard that encourages the use of 4 drugs, all subjects -both in active comparator and experimental arm- will also receive isoniazide 300 mg p.o. and pyrazinamide 1500 mg p.o.
  Unconscious subjects will receive oral drugs via nasogastric tubes (NGT)
  Interventions: Drug: Moxifloxacin
- High dose rifampisin (Experimental): Subjects in this arm receive 600 mg Rifampisin i.v. for 14 days, and the dosage will be switched to 450 mg Rifampisin p.o afterwards until completion of TB medication (in accordance with National TB Program)
  In accordance with national TB treatment standard that encourages the use of 4 drugs, all subjects -both in active comparator and experimental arm- will also receive isoniazide 300 mg p.o. and pyrazinamide 1500 mg p.o.
  Unconscious subjects will receive oral drugs via nasogastric tubes (NGT)
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Moxifloxacin — Subjects on both arms will further be randomized into receiving moxifloxacin either in standard dose (400 mg p.o.), high dose (800 mg p.o.) of moxifloxacin, or not receiving moxifloxacin (ethambutol 750 mg p.o., instead) Intervention drug will be given for 14 days, and the drug will be switched to ethambutol 750 mg p.o. (in accordance with National TB Program)
  Other Names: Avelox (r)

SUMMARY:
Tuberculous meningitis (TBM) is the most lethal form of tuberculosis infection, and is diagnosed in approximately 5-10% of TB patients. The incidence of TBM has increased considerably during the last decade, partly due to the HIV epidemic. Without treatment, virtually all patients with TB meningitis will die. With the current treatment regimens, TBM is fatal in approximately 30-50% of cases, and responsible for severe disability in a similar proportion of survivors.

Worldwide, Indonesia the third highest case load of tuberculosis with an estimated 500,000 new patients / year. Representative data are lacking, but it is clear that TBM is a growing problem. For instance, in Hasan Sadikin Hospital, the top-referral hospital for West Java Province (population 40 million), Indonesia, 40-50 cases of TBM were treated yearly in the late 90's compared to approximately 100 in recent years.

There is very little evidence for the current treatment regimen for TBM, which dates back to the late 60's. Therefore, there is an urgent need to evaluate intensified treatment of TBM in randomized trials. We hypothesize that higher dose rifampicin, moxifloxacin (possibly also at high dose), or both will improve outcome of TBM. To determine the experimental regimen(s) which should be compared with current regimen in phase 3 trials, we want to evaluate pharmacokinetic aspects and toxicity of candidate regimens in a phase 2 clinical trial in 60 patients with TBM in Indonesia.

ELIGIBILITY:
Inclusion Criteria:

* Tuberculous meningitis, diagnosed based on clinical and/or CSF criteria
* Age 15 years old or more
* Hospitalized for the treatment

Exclusion Criteria:

* Pregnancy/lactation
* On TB treatment within 7 days before inclusion
* Elevated liver enzyme (> 5x than normal values)
* Known hypersensitivity/intolerance to rifampicin or moxifloxacin
* Prolonged QTc interval in ECG or other detectable cardiac arrythmias, in the absence of hypokalemia
* Refusal to be included in the study

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Rifampicin and Moxifloxacin concentration in plasma and CSF | Plasma drug concentration samplings at 0, 1, 2, 4, 6 and 24h post dose (6 time points). CSF samples at 2 time points.
  On sampling day (one of the first 3 days of hospitalization), we will measure plasma and CSF drug concentration at several time points.
  Plasma drug concentration will be measured at 6 time points (hour 0, 1, 2, 4, 6 and 12).
  CSF drug concentration at 2 time points: (1) hour 3-6 post dose on the same blood sampling day and (2) within 5 days after the 1st day of TB drug administration, 1-3 hours after drug intake

SECONDARY OUTCOMES:
Early and late mortality | 1st and 6th month of TB treatment
  We will measure early (within first month of TB treatment) and late (after 6 months of TB treatment) mortality

CONTACTS AND LOCATIONS:
Overall Officials: Rovina Ruslami, PhD, Principal Investigator — Faculty of Medicine, Universitas Padjadjaran, Bandung, Indonesia
Locations (1):
- Hasan Sadikin General Hospital, Bandung, West Java, Indonesia

REFERENCES:
- [Derived] Te Brake L, Dian S, Ganiem AR, Ruesen C, Burger D, Donders R, Ruslami R, van Crevel R, Aarnoutse R. Pharmacokinetic/pharmacodynamic analysis of an intensified regimen containing rifampicin and moxifloxacin for tuberculous meningitis. Int J Antimicrob Agents. 2015 May;45(5):496-503. doi: 10.1016/j.ijantimicag.2014.12.027. Epub 2015 Feb 7. PMID 25703312
- [Derived] Ruslami R, Ganiem AR, Dian S, Apriani L, Achmad TH, van der Ven AJ, Borm G, Aarnoutse RE, van Crevel R. Intensified regimen containing rifampicin and moxifloxacin for tuberculous meningitis: an open-label, randomised controlled phase 2 trial. Lancet Infect Dis. 2013 Jan;13(1):27-35. doi: 10.1016/S1473-3099(12)70264-5. Epub 2012 Oct 25. PMID 23103177